CLINICAL TRIAL: NCT01431716
Title: A Multicenter, Single-arm, Open-label, Phase 3b Study to Assess the Effects of Switching From Flolan® to EFI/ACT-385781A in Patients With Pulmonary Arterial Hypertension
Brief Title: Epoprostenol for Injection (EFI/ACT-385781A) - Pulmonary Arterial Hypertension
Acronym: EPITOME-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-066A301
Record Dates: First submitted 2011-09-07; First posted 2011-09-12 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Epoprostenol; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EFI/ACT-385781A (Experimental): EFI/ACT-385781 administered by continuous intravenous infusion via a central venous catheter using an ambulatory infusion pump
  Interventions: Drug: EFI/ACT-385781A

INTERVENTIONS:
Drug: EFI/ACT-385781A
  Other Names: ACT-385781A; Epoprostenol for injection (EFI)

SUMMARY:
This study is investigating the effect of switching from Flolan® to Epoprostenol for Injection (EFI/ACT-385781A) in pulmonary arterial hypertension patients currently treated with Flolan®. For this purpose patients being treated for at least 12 months with Flolan® will be switched from Flolan® to EFI/ACT-385781A and followed-up for 90 days. During these 90 days safety and tolerability of EFI/ACT-385781A will closely be monitored in all treated patients. This 90 follow-up will provide clinical evidence on the safety, tolerability, efficacy and treatment satisfaction of switching from Flolan® to EFI/ACT-385781A in patients with pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years and above
2. Patients with the following types of pulmonary arterial hypertension (PAH) belonging to WHO Group I: Idiopathic (IPAH), Heritable (HPAH), Associated (APAH) with Connective tissue diseases or Drugs and toxins
3. Patients treated with Flolan® for at least 12 months and on a stable dose for at least 3 months prior to enrollment
4. Patients who are currently treated with concomitant PAH therapy listed below must have been treated for at least 90 days and on a stable dose for 30 days prior to enrollment: Bosentan, Ambrisentan, Sitaxsentan, Sildenafil, Tadalafil
5. Women of childbearing potential must use a reliable method of contraception
6. Signed informed consent prior to initiation of any study mandated procedure

Exclusion Criteria:

1. Patients with respiratory and/or cardiovascular distress in need of emergency care
2. Known or suspicion of pulmonary veno-occlusive disease (PVOD)
3. Current use of IV inotropic agents
4. Current use of any prostacyclin or prostacyclin analog other than Flolan®
5. Tachycardia with heart rate > 120 beats/min at rest
6. PAH related to any condition other than those specified in the inclusion criteria
7. Known hypersensitivity to the formulations EFI/ACT-385781A or any of its excipients, and Flolan® or any of its excipients
8. Cerebrovascular events (e.g., transient ischemic attack or stroke) within 6 months of screening
9. History of myocardial infarction
10. History of left-sided heart disease, including any of the following:

    * hemodynamically significant aortic or mitral valve disease
    * restrictive or congestive cardiomyopathy
    * left ventricular ejection fraction < 40% by multigated radionucleotide angiogram (MUGA), angiography, or echocardiography
    * unstable angina pectoris
    * life-threatening cardiac arrhythmias
11. Chronic bleeding disorders
12. Central venous line infection within 90 days prior to screening and/or a history of recurring line infections
13. Women who are pregnant or breast-feeding
14. Participation in another clinical trial, except observational, or receipt of an investigational product within 30 days prior to randomization
15. Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence or psychiatric disease
16. Known concomitant life-threatening disease other than PAH with a life expectancy < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- UZ Gasthuisberg, Leuven, Belgium
- Canada (2):
  - University Health Network, Toronto TGH - 10 EN - 220, Toronto, Ontario
  - Sir Mortimer B Davis Jewish General Hospital, Montreal, Quebec
- France (2):
  - Centre Hospitalier Universitaire, Caen
  - Hôpital Antoine Béclère, Clamart
- Orsola Malpighi, Bologna, Italy
- VU Medisch Centrum (VUMC), Amsterdam, Netherlands
- Hospital Vall d'Hebron, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at eight centers in the European Union and Canada. First patient, first visit was 15 March 2011 and last patient, last visit was 2 February 2012.
Pre-assignment Details: Patients must have been treated with Flolan for at least 12 months and on a stable dose for at least 3 months prior to enrollment. There was a screening period of up to 14 days.
Groups:
- Epoprostenol for Injection (EFI/ACT-385781A): EFI/ACT-385781A administered by continuous intravenous infusion via a central venous catheter using an ambulatory infusion pump.
Period: Overall Study
Arm/Group | Epoprostenol for Injection (EFI/ACT-385781A)
Started | 42
Completed | 41
Not Completed | 1
Not completed — Withdrawal of consent | 1

BASELINE CHARACTERISTICS:
Population: All-treated set (One patient enrolled in the study but withdrew consent prior completing baseline assessment and receiving study drug).
Groups:
- EFI/ACT-385781A: EFI/ACT-385781A administered by continuous intravenous infusion via a central venous catheter using an ambulatory infusion pump.
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (13.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 11
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 18
  Black | 2
  Asian | 1
  Not Collected | 20
Region of Enrollment [Number; unit: participants]
  France | 20
  Canada | 8
  Spain | 2
  Belgium | 5
  Netherlands | 4
  Italy | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Vascular Resistance From Baseline to End of Treatment (EOT).
Description: Right heart catheterization was performed for cardiac hemodynamic assessment at Screening or Day 1, prior to switch from Flolan® to EFI/ACT-385781A and at EOT.
Time Frame: Approximately 3 months
Population: All treated set without imputation for missing values. Data was missing for 5 patients.
Measure: Mean (Standard Deviation); unit: dyn/sec/cm^5
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 36
dyn/sec/cm^5
  Baseline | 595.70 (237.14)
  End of treatment | 587.66 (248.44)

2. Other Pre Specified Outcome: Change in 6-minute Walk Distance (6MWD) From Baseline to EOT.
Description: The 6MWD was assessed at Screening or Day 1, prior to switch from Flolan® to EFI/ACT-385781A and at EOT. The 6-minute walk test is a non-encouraged test that measures the distance walked for the duration of 6 min.
Time Frame: Approximately 3 months
Population: All-treated set who had both a baseline and an EOT assessment.
Measure: Mean (Standard Deviation); unit: m
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 40
m
  Baseline | 498.1 (86.0)
  End of treatment | 492.8 (81.6)

3. Primary Outcome: Change in Total Pulmonary Resistance From Baseline to End of Treatment (EOT).
Description: as for outcome 1
Time Frame: Approximately 3 months
Population: All treated set without imputation for missing values
Measure: Mean (Standard Deviation); unit: dyn/sec/cm^5
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 41
dyn/sec/cm^5
  Baseline | 752.44 (260.91)
  End of treatment | 757.51 (296.82)

4. Primary Outcome: Change in Mean Pulmonary Arterial Pressure From Baseline to End of Treatment (EOT).
Description: as for outcome 1
Time Frame: Approximately 3 months
Population: All treated set without imputation for missing values
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 41
mmHg
  Baseline | 51.9 (11.5)
  End of treatment | 51.7 (12.8)

5. Primary Outcome: Change in Mean Right Atrial Pressure From Baseline to End of Treatment (EOT).
Description: as for outcome 1
Time Frame: Approximately 3 months
Population: All treated set without imputation for missing values
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 41
mmHg
  Baseline | 7.9 (4.6)
  End of treatment | 7.1 (4.6)

6. Primary Outcome: Change in Pulmonary Capillary Wedge Pressure From Baseline to End of Treatment (EOT).
Description: as for outcome 1
Time Frame: Approximately 3 months
Population: All treated set without imputation for missing values. Data was missing for 5 patients.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 36
mmHg
  Baseline | 10.3 (3.8)
  End of treatment | 10.1 (4.3)

7. Primary Outcome: Change in Mean Cardiac Index From Baseline to End of Treatment (EOT).
Description: as for outcome 1
Time Frame: Approximately 3 months
Population: All treated set without imputation for missing values
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 41
L/min/m^2
  Baseline | 3.34 (0.71)
  End of treatment | 3.38 (0.81)

8. Other Pre Specified Outcome: Change in Borg Dyspnea Score From Baseline to EOT.
Description: The Borg dyspnea score was assessed at Screening or Day 1, prior to switch from Flolan® to EFI/ACT-385781A and at EOT. The Borg scale is a category-ratio scale, commonly used to evaluate the effects of exercise on dyspnea. The original and modified scales have ratio properties ranging from 0 = nothing at all to 10 = very, very severe, with descriptors from 0 to 10. Descriptors have been modified by others so that 10 has been labelled "extremely severe," or "the worst possible dyspnea imaginable."
Time Frame: Approximately 3 months
Population: All-treated set who had both a baseline and an EOT assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 40
units on a scale
  Baseline | 4.0 (2.1)
  End of treatment | 3.3 (2.1)

9. Other Pre Specified Outcome: Number of Participants With Improved, No Change, or Worsening of New York Heart Association Functional Class (NYHA FC) From Baseline to EOT.
Description: NYHA FC was assessed at Screening or Day 1, prior to switch from Flolan® to EFI/ACT-385781A and at EOT. Disease severity was assessed by NYHA classification of pulmonary arterial hypertension criteria: Class I: no limitation of physical activity (PA). Ordinary PA: no undue dyspnea/fatigue, chest pain, near syncope. Class II: slight limitation of PA. Comfortable at rest. Ordinary PA: undue dyspnea/fatigue, chest pain, near syncope. Class III: marked limitation of PA. Comfortable at rest. Less than ordinary PA: undue dyspnea/fatigue, chest pain, near syncope. Class IV: inability to carry out PA without symptoms. Right heart failure. Dyspnea/fatigue may even have been present at rest. Discomfort increased by any PA.
Time Frame: Approximately 3 months
Population: All-treated set who had both a baseline and an EOT assessment.
Measure: Number; unit: participants
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 40
participants
  Improved | 1
  No change | 35
  Worsened | 4

10. Other Pre Specified Outcome: Change in N-terminal Pro-B-type Natriuretic Peptide (NT proBNP) From Baseline to EOT.
Description: Blood sampling for NT proBNP was performed at Screening or Day 1, prior to switch from Flolan® to EFI/ACT-385781A and at EOT.
Time Frame: Approximately 3 months
Population: All-treated set who had both a baseline and an EOT assessment.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 36
ng/L
  Baseline | 599.97 (1164.21)
  End of treatment | 613.56 (1155.90)

11. Other Pre Specified Outcome: Change in Effectiveness Score of the Abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9) From Baseline to EOT.
Description: Patients were required to complete the TSQM-9 questionnaire at Screening or Day 1, prior to switch from Flolan® to EFI/ACT-385781A and at EOT. The TSQM-9 is a validated instrument to assess patients' satisfaction with medication, including a three question effectiveness scale. The TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain.
Time Frame: Approximately 3 months
Population: All-treated set who had both a baseline and an EOT assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 38
units on a scale
  Baseline | 78.22 (12.61)
  End of treatment | 74.71 (17.60)

12. Other Pre Specified Outcome: Change in Convenience Score of the Abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9) From Baseline to EOT.
Description: Patients were required to complete the TSQM-9 questionnaire at Screening or Day 1, prior to switch from Flolan® to EFI/ACT-385781A and at EOT. The TSQM-9 is a validated instrument to assess patients' satisfaction with medication, including a three question convenience scale. The TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain.
Time Frame: Approximately 3 months
Population: All-treated set who had both a baseline and an EOT assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 38
units on a scale
  Baseline | 53.65 (15.78)
  End of treatment | 66.37 (17.04)

13. Other Pre Specified Outcome: Change in Global Satisfaction Score of the Abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9) From Baseline to EOT.
Description: Patients were required to complete the TSQM-9 questionnaire at Screening or Day 1, prior to switch from Flolan® to EFI/ACT-385781A and at EOT. The TSQM-9 is a validated instrument to assess patients' satisfaction with medication, including a three question global satisfaction scale. The TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain.
Time Frame: Approximately 3 months
Population: All-treated set who had both a baseline and an EOT assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 38
units on a scale
  Baseline | 71.82 (18.35)
  End of treatment | 75.22 (15.58)

14. Other Pre Specified Outcome: Number of Participants With Adverse Events Leading to Discontinuation of Study Drug From Baseline to EOT.
Description: Adverse events that led to discontinuation of study drug from the start of study treatment until the end of study treatment were recorded.
Time Frame: Approximately 3 months
Population: All-treated set.
Measure: Number; unit: participants
Arm/Group | EFI/ACT-385781A
Number analyzed (Participants) | 41
participants | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) that occurred from the start of study treatment until 24 h after the end of study treatment were recorded. In addition, all serious AEs that occurred up to 30 days after the end of study treatment were also recorded.
Description: All treated set
Arm/Group | EFI/ACT-385781A
Serious Adverse Events (participants affected / at risk) | 7/41
Other Adverse Events (participants affected / at risk) | 31/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EFI/ACT-385781A (N=41)
Diverticulitis (Infections and infestations) | 1
Device-related infection (pseudomonas) (Infections and infestations) | 1
Device connection issue (General disorders) | 2
Right ventricular failure (Cardiac disorders) | 1
Device damage (General disorders) | 1
Device dislocation (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EFI/ACT-385781A (N=41)
HEADACHE (Nervous system disorders) | 12
NASOPHARYNGITIS (Infections and infestations) | 7
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 6
FLUSHING (Vascular disorders) | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3
PALPITATIONS (Cardiac disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less